CLINICAL TRIAL: NCT00206427
Title: A Neoadjuvant Phase II Trial of GW572016 in HER2 Overexpressing Breast Cancer Patients: Biologic Correlative Study
Brief Title: Neoadjuvant GW572016 to Treat Breast Cancer
Acronym: GW
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Baylor Breast Care Center (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Mothaffar Rimawi, Medical Director, Baylor Breast Care Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H 15430; Neoadjuvant GW572016 (Other: Baylor Breast Center)
Record Dates: First submitted 2005-09-14; First posted 2005-09-21 (Estimated); Results first posted 2012-03-07 (Estimated); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Breast Cancer
Keywords: Advanced; Breast; Cancer; Neoadjuvant; HER2
MeSH Terms: conditions — Breast Neoplasms; Neoplasms | interventions — Lapatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intervention (Experimental): Intervention/Lapatinib (GW572016)
  Interventions: Drug: GW572016; Drug: lapatinib

INTERVENTIONS:
Drug: GW572016 — Lapatinib, 500 mg
  Other Names: TyKerb; Lapatinib
Drug: lapatinib — Lapatinib 500 mg PO
  Other Names: TyKerb; GW572016

SUMMARY:
We want to learn whether GW572016 is effective in breast cancers that have HER2.

DETAILED DESCRIPTION:
The EGFR/HER family of transmembrane type I receptor tyrosine kinases are enzymes that play an important role in fundamental cell processes like cell proliferation, differentiation, and survival. These receptor tyrosine kinases, which include HER1 (epidermal growth factor receptor, EGFR), HER2 (HER2/neu, c-erbB2), HER3 and HER4 contain an extracellular domain and intracellular protein tyrosine kinase core. Aberrant HER1 and HER2 signaling has been causally associated with cancer cell proliferation and survival.

HER1 is expressed or over-expressed in many human solid tumors and plays an important role in progression to invasion and metastases.. The association between HER2 overexpression and poor prognosis in node-positive and advanced breast cancer has been shown by a number of studies. Based on this association between the members of HER1/HER2 family and worse clinical outcome, antibodies and small molecules that specifically target these receptor tyrosine kinases were developed for their therapeutic efficacy.

Trastuzumab (Herceptin) is a highly purified recombinant DNA-derived humanized monoclonal antibody that selectively binds with high affinity to the extracellular domain of the HER2 receptor. Pivotal multicenter efficacy trials in metastatic patients showed improved response rates and disease-free survival in patients who received trastuzumab in addition to chemotherapy. One of these studies was an open-labeled, multicenter, randomized phase III study evaluating the addition of trastuzumab to standard first-line chemotherapy in metastatic breast cancer. This study randomized 469 patients with metastatic disease to chemotherapy with or without trastuzumab. Results of this study showed survival in patients who received trastuzumab plus chemotherapy to be almost twice as long as chemotherapy alone (7.2 vs. 4.5 months, p<0.0001).

As dimerization is important in signal transduction, therapies that target more than one member of the HER family may have greater anti-tumor effect. Recently, data with trastuzumab plus IMC-C224 in human ovarian cancer cells showed greater growth inhibition compared to either monoclonal antibody alone. GW572016 is an orally active dual HER1/HER2 kinase inhibitor that blocks signal transduction pathways. This dual inhibition is an attractive therapeutic strategy for epithelial cancers, as ligand-induced HER1/HER2 dimerization triggers off potent proliferative and survival signals. In vitro studies with GW572016 have shown marked activity, leading to growth arrest and apoptosis in HER1 and HER2 overexpressing cell lines. GW572016 markedly reduced tyrosine phosphorylation of HER1 and HER2, and activation of MAP kinase and Akt, the downstream effectors of proliferation and survival, respectively. In vitro studies in HER-2 overexpressing cell lines have demonstrated synergistic activity when GW572016 is combined with taxanes. Phase I studies with GW572016 and taxanes have been completed, with results demonstrating that this small molecule inhibitor may be safely combined with chemotherapy with no unanticipated side effects.

The EGFR/HER family of transmembrane type I receptor tyrosine kinases are enzymes that play an important role in fundamental cell processes like cell proliferation, differentiation, and survival. These receptor tyrosine kinases, which include HER1 (epidermal growth factor receptor, EGFR), HER2 (HER2/neu, c-erbB2), HER3 and HER4 contain an extracellular domain and intracellular protein tyrosine kinase core. Aberrant HER1 and HER2 signaling has been causally associated with cancer cell proliferation and survival.

Trastuzumab (Herceptin) is a highly purified recombinant DNA-derived humanized monoclonal antibody that selectively binds with high affinity to the extracellular domain of the HER2 receptor. Results of this study showed survival in patients who received trastuzumab plus chemotherapy to be almost twice as long as chemotherapy alone (7.2 vs. 4.5 months, p<0.0001).

In vitro studies with GW572016 have shown marked activity, leading to growth arrest and apoptosis in HER1 and HER2 overexpressing cell lines. GW572016 markedly reduced tyrosine phosphorylation of HER1 and HER2, and activation of MAP kinase and Akt, the downstream effectors of proliferation and survival, respectively. In vitro studies in HER-2 overexpressing cell lines have demonstrated synergistic activity when GW572016 is combined with taxanes. Phase I studies with GW572016 and taxanes have been completed, with results demonstrating that this small molecule inhibitor may be safely combined with chemotherapy with no unanticipated side effects.

As the type I tyrosine kinases are involved in various aspects of cell growth and survival, a potent quinazoline and pyrido-[3,4-d]-pyrimidine small molecule (GW572016) against HER1 and HER2 was developed which showed potent in vitro inhibition of HER1 and HER2 in tumor cell lines. Mouse xenograft models of BT474 and HN5 cell lines also showed growth inhibition in a dose-responsive manner. In addition, GW572016 caused a reduction in HER1 and HER2 autophosphorylation, indicating interference of this signaling pathway. GW572016 not only inhibited baseline activation of HER1 and HER2, but also has been shown to interrupt downstream activation of Erk1/2 MAP kinases and Akt.

HER1 is expressed or over-expressed in many human solid tumors and plays an important role in progression to invasion and metastases.. The association between HER2 overexpression and poor prognosis in node-positive and advanced breast cancer has been shown by a number of studies. Based on this association between the members of HER1/HER2 family and worse clinical outcome, antibodies and small molecules that specifically target these receptor tyrosine kinases were developed for their therapeutic efficacy.

Trastuzumab (Herceptin) is a highly purified recombinant DNA-derived humanized monoclonal antibody that selectively binds with high affinity to the extracellular domain of the HER2 receptor. Pivotal multicenter efficacy trials in metastatic patients showed improved response rates and disease-free survival in patients who received trastuzumab in addition to chemotherapy. One of these studies was an open-labeled, multicenter, randomized phase III study evaluating the addition of trastuzumab to standard first-line chemotherapy in metastatic breast cancer. This study randomized 469 patients with metastatic disease to chemotherapy with or without trastuzumab. Results of this study showed survival in patients who received trastuzumab plus chemotherapy to be almost twice as long as chemotherapy alone (7.2 vs. 4.5 months, p<0.0001).

We have completed the first single-agent neoadjuvant trastuzumab study in human breast cancer. The specific aims of this study were to firstly, define the clinical efficacy of trastuzumab, and secondly, to determine its mechanism of action in human breast cancer specimens. From September 1999 to June 2003, 27 patients with HER2 overexpressing locally advanced breast cancer with or without gross metastatic disease, were considered for a phase II study with neoadjuvant trastuzumab. At presentation, the median tumor size was large at 8x8 cm2 (range 4x4 cm2 to 25x20 cm2). We did not expect measurable evidence of tumor regression with this short treatment duration. However, regression in the product of bidimensional tumor measurements with a median decrease of -20.0% (range 0, -60.4%, p=0.0001) was observed in primary tumors after only 3 weeks of single agent trastuzumab. Most surprisingly, partial response was observed in 26% (7/27). Minor response was seen in 44% (12/27), and stable disease in 30% (8/27). No tumors increased in size during this 3-week period.

This is the first neoadjuvant trastuzumab monotherapy study in treatment-naive patients with HER2 overexpressing breast cancers. The clinical efficacy with tumor reductions in some patients presenting with large initial tumors indicates that the monoclonal antibody can be safely administered as a single agent without fear of tumor progression. When the study was first started, the uncertainty of the clinical efficacy of neoadjuvant single agent trastuzumab limited its duration to 3 weeks. It seems likely that the true response rate would have been higher if therapy was continued for several months. Based on these data, longer treatment durations of HER2 targeted therapy, like with GW572016, given as a single agent should be investigated in clinical trials with careful monitoring of patients to assess its activity in this setting.

Aim 1: To demonstrate the clinical efficacy of GW572016 when given as neoadjuvant therapy as a single agent in patients with treatment-naive, locally advanced HER2 overexpressing breast cancer. We aim to discover the true response rate to inhibiting HER1/2 signal transduction with GW572016 in breast cancer patients.

Aim 2: To determine if GW572016 inhibits HER1 and HER2 signaling in situ.The mechanism of therapeutic action of GW572016 is not fully understood.

ELIGIBILITY:
Inclusion Criteria:

1. All patients must be female.
2. Signed informed consent.
3. Locally advanced breast cancers or primary breast cancers with concomitant gross metastatic disease are eligible. Locally advanced cancers must be of clinical and/or radiologic size >/- 5 cm, and/or are deemed surgically inoperable, with Stage IIIb, IIIc, or IV disease.
4. HER2 overexpressing tumors defined as HercepTest score of 3+, or >/- 10% cells moderately or strongly HER2 positive by other methods, or semi-quantitative score of >/- 5 (in Dr. Allred's laboratory) or gene amplified.
5. Negative serum pregnancy test (BHCG) within 7 days of starting study, if of child-bearing potential.
6. Kidney and liver function tests - all within 1.5 times the institution's upper limit of normal.
7. Performance status (WHO scale) less than 2 and life expectancy greater than 6 months.
8. Age greater than 18 years.
9. No brain or leptomeningeal disease.
10. No previous or current malignancies at other sites within the last 5 years, with exception of adequately treated core-biopsied in situ carcinoma of the cervix uteri and basal or squamous cell carcinoma of the skin.

Exclusion Criteria:

1. Pregnancy or unwillingness to use a reliable contraceptive method in women of child-bearing potential.
2. Severe underlying chronic illness or disease.
3. Cardiomyopathy or baseline LVEF <50%.
4. Other investigational drugs while on study.
5. Severe or uncontrolled hypertension, history of congestive heart failure or severe coronary arterial disease.
6. Malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel. Subjects with ulcerative colitis are also excluded.
7. Taking any GW572016-prohibited medication (see GW572016 Prohibited Medications List in protocol) within 7 days of first dose of study medications.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2004-08; Primary Completion 2011-06 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mothaffar Rimawi, MD, Principal Investigator — Baylor Breast Center
Locations (3):
- United States (3):
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - University of New Mexico, Albuquerque, New Mexico
  - Baylor Breast Center, Houston, Texas

REFERENCES:
- See also: Web site — http://www.breastcenter.tmc.edu

RESULTS

PARTICIPANT FLOW:
Groups:
- GW572016 1500mg: The study had only 1 treatment group and all patient had GW572016 1500mg daily.
Period: Overall Study
Arm/Group | GW572016 1500mg
Started | 49 (Received First Dose)
Completed | 47 (Complete 6-week therapy)
Not Completed | 2
Not completed — Adverse Event | 2

BASELINE CHARACTERISTICS:
Groups:
- GW572016 1500mg: patients received GW572016 1500mg daily
Arm/Group | GW572016 1500mg
Number analyzed (Participants) | 49
Age, Continuous [Median (Full Range); unit: years] | 53 [27 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Clinical Response
Description: Clinical efficacy was assessed by bidimensional tumor measurements of the primary cancer at baseline, and at the end of week 6. Clinical complete response (cCR) was defined as complete disappearance of the primary tumor. Clinical partial response (cPR) was defined as a decrease by at least 50% of the sum of the products of the largest perpendicular diameters. An increase of more than 25% was defined as clinical progressive disease (cPD). Any response that does not meet the definition of cCR, cPR, or cPD was defined as stable disease (cSD).
Time Frame: at the end of week 6.
Population: All patients finished 6-week therapy were included. Two patients dropped off therapy early were excluded.
Measure: Number; unit: participants
Arm/Group | GW572016 1500mg
Number analyzed (Participants) | 47
participants
  cCR | 3
  cPR | 30
  cSD | 11
  cPD | 3

2. Secondary Outcome: Inhibition of HER1 and HER2 Signaling as Determined by EGFR, HER2, and pHER2
Description: Immunohistochemical staining of cells from patients breast biopsies at baseline and post-treatment (week 6) were performed. Biologic markers including EGFR, HER2, and pHER2 were assessed with intensity scores of the staining (0-3, higher score means higher intensity).
Time Frame: Baseline and 6 weeks
Population: Samples from 47 patients who finished 6-week therapy were included. The numbers of biomarker data depended on available data due to missed biopsies or no tumor found in some samples.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | GW572016 1500mg
Number analyzed (Participants) | 47
score on a scale
  EGFR at baseline: number analyzed (Participants) | 35
  EGFR at baseline | 0 [0 to 1]
  EGFR at week 6: number analyzed (Participants) | 21
  EGFR at week 6 | 0 [0 to 1]
  HER2 at baseline: number analyzed (Participants) | 36
  HER2 at baseline | 3 [2.75 to 3]
  HER2 at week 6: number analyzed (Participants) | 28
  HER2 at week 6 | 3 [2.5 to 3]
  pHER2 at baseline: number analyzed (Participants) | 36
  pHER2 at baseline | 1.5 [0 to 2.5]
  pHER2 at week 6: number analyzed (Participants) | 24
  pHER2 at week 6 | 1.5 [0 to 2.5]

3. Secondary Outcome: Inhibition of HER1 and HER2 Signaling as Determined by ki67 and CC3
Description: Immunohistochemical staining of cells from patients breast biopsies at baseline and post-treatment (week 6) were performed. Biologic markers of Ki67 and CC3 were assessed with percentages of cells staining positive (0%-100%, higher score means higher positive cells).
Time Frame: Baseline and 6 weeks
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: percentage of cells staining positive
Arm/Group | GW572016 1500mg
Number analyzed (Participants) | 47
percentage of cells staining positive
  Ki67 at baseline: number analyzed (Participants) | 34
  Ki67 at baseline | 71 [54 to 78]
  Ki67 at week 6: number analyzed (Participants) | 22
  Ki67 at week 6 | 49 [29 to 65]
  CC3 at baseline: number analyzed (Participants) | 35
  CC3 at baseline | 1.80 [0.82 to 3.11]
  CC3 at week 6: number analyzed (Participants) | 21
  CC3 at week 6 | 1.84 [0.50 to 5.31]

ADVERSE EVENTS:
Time Frame: During the 6-week therapy
Arm/Group | GW572016 1500mg
Serious Adverse Events (participants affected / at risk) | 3/49
Other Adverse Events (participants affected / at risk) | 32/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GW572016 1500mg (N=49)
rash (Skin and subcutaneous tissue disorders) | 1 (1)
Neutrophils/ANC (Blood and lymphatic system disorders) | 1 (2)
Leukocytes (Blood and lymphatic system disorders) | 1 (3)
Hypocalcemia (Blood and lymphatic system disorders) | 1 (5)
Constipation (Gastrointestinal disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Infection-oral thrush (Infections and infestations) | 1 (2)
Mucositis-oral (Gastrointestinal disorders) | 1 (2)
Left Ventricular Systolic Dysfunction (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GW572016 1500mg (N=49)
Bruising (Skin and subcutaneous tissue disorders) | 3 (4)
Diarrhea (Gastrointestinal disorders) | 23 (26)
Elevated AST (Hepatobiliary disorders) | 4 (4)
Nausea (Gastrointestinal disorders) | 4 (4)
Pruritis (Skin and subcutaneous tissue disorders) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 18 (20)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes